CLINICAL TRIAL: NCT04883034
Title: Adductor Canal Block in Outpatient Clinic
Brief Title: Adductor Canal Block in Outpatient Clinic for Pain Control After Knee Arthroplasty
Acronym: ACB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Sholahuddin Rhatomy, Head Of orthopaedic and Traumatology Department, Dr Soeradji Tirtonegoro Hospital/Faculty of Medicine, Public Health and Nursing, Universitas Gadjah Mada, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACB OUTPATIENT CLINIC
Record Dates: First submitted 2021-04-30; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Acute Pain; Total Knee Arthroplasty
MeSH Terms: conditions — Acute Pain | interventions — Ambulatory Care Facilities; Analgesics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pain management post total knee arthroplasty with analgetic oral (Placebo Comparator): Patients in control group were given analgesic (etoricoxibe) on a daily basis, with the option to increase the dose if pain persisted, up to a maximum of 120 mg per day.
  Interventions: Drug: Analgesics, etoricoxibe
- pain management post total knee arthroplasty with adductor canal block (Active Comparator): On postoperative day 14 (POD 14), the ACB was performed for ACB group
  Interventions: Procedure: adductor canal block in outpatient clinic

INTERVENTIONS:
Procedure: adductor canal block in outpatient clinic — perform adductor canal block in outpatient clinic for patient post total knee arthroplasty
  Arms: pain management post total knee arthroplasty with adductor canal block
Drug: Analgesics, etoricoxibe — anaelgetic oral intake
  Other Names: etoricoxibe
  Arms: pain management post total knee arthroplasty with analgetic oral

SUMMARY:
Single-shot Adductor Canal Block in the outpatient clinic is safe, significantly decreased pain and analgesic consumption and may enhance the rehabilitation program

DETAILED DESCRIPTION:
The ACB in the outpatient clinic is safe and can minimize postoperative pain. The primary goal of this research was to see how ACB affected the Visual Analog Score (VAS) pain score during the rehabilitation as opposed to controls. The secondary goal was to determine how much analgesic (etoricoxibe) was consumed on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Indonesian or Javanese-speaking adults
* After perfomed total knee replacement
* American Society of Anesthesiologists physical status I-III
* body mass index (BMI) of 18-40 kg/m2

Exclusion Criteria:

* Declined to complete the study
* Unable to cooperate
* had an allergic reaction to any of the drugs
* abusing alcohol or drugs

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog pain score (VAS) | one month
  A VAS scale was used to assess pain severity, with 0 indicating no pain and 10 indicating extreme pain

SECONDARY OUTCOMES:
analgesic oral intake (etoricoxibe) | one month
  determine how much analgesic (etoricoxibe) was consumed on a daily basis.

CONTACTS AND LOCATIONS:
Overall Officials: sholahuddin rhatomy, dr, Principal Investigator — Gadjah Mada University
Locations (1):
- Sholahuddin Rhatomy, Sleman, Special Region of Yogyakarta, Indonesia